CLINICAL TRIAL: NCT05284461
Title: Effect of Shape and Surface Treatment of the Transmucosal Abutments on the Bone-implant-contact and the Peri-implant Health, .
Brief Title: Effect of Shape and Surface Treatment of the Transmucosal Abutments on Peri-implant Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Professor in Prosthodontics, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USAL_2021_JMONT
Record Dates: First submitted 2022-02-02; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Edentulous; Alveolar Process, Atrophy
MeSH Terms: conditions — Mouth, Edentulous; Atrophy | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mechanized parallel abutments (Placebo Comparator): Implants were immediately covered with this type of abutments after insertion. This is the most common procedure. It would be the gold standard
  Interventions: Device: dental implant with transepithelial abutments manufactured by Galimplant Dental System (Spain)
- Anodized parallel abutments (Experimental): Implants were immediately covered with this kind of abutments after insertion. Only the surface treatment varies to the gold standard
  Interventions: Device: dental implant with transepithelial abutments manufactured by Galimplant Dental System (Spain)
- Mechanized convergent abutments (Experimental): Implants were immediately covered with this kind of abutments after insertion. Only the geometry of the emergence profile varies with regards to the gold standard
  Interventions: Device: dental implant with transepithelial abutments manufactured by Galimplant Dental System (Spain)
- Anodized convergent abutments (Experimental): Implants were immediately covered with this kind of abutments after insertion. Both the surface treatment and the geometry vary with regards to the gold standard
  Interventions: Device: dental implant with transepithelial abutments manufactured by Galimplant Dental System (Spain)

INTERVENTIONS:
Device: dental implant with transepithelial abutments manufactured by Galimplant Dental System (Spain) — Dental implants with transepithelial abutments with distinct morphology

SUMMARY:
The sample was comprised by 10 patients in which 40 dental implants are placed in an atrophic maxilla. All the implants were connected to 4 types of transepithelial abutment: i.e: parallel anodized abutment(n=10); parallel mechanized abutmen(n=10)t, convergent anodized abutment(n=10); and convergent mechanized abutment (n=10) three months after insertion implants were extracted with the surrounding hard and soft tissues for the histological evaluation of the clinical performance.

ELIGIBILITY:
Inclusion Criteria:

* totally edentulous patients in the upper arch and carriers of conventional complete dentures for more than ten years, without temporomandibular disorders

Exclusion Criteria:

* evidence of systemic or psychic pathology that contraindicates implant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Bone to implant contact | 3 months after healing
  It is a Percentage estimation of native bone in direct contact to implant determined by histological assessments (optical microscopy)
Peri-implant inflammation of the soft tissues | 3 months after healing
  Histological assessments as ordinal variables of the grade of inflammatory infiltrate (none, minor, major)according to standard guidelines.
Density of the peri-implant soft tissues | 3 months after healing
  Histological assessments as ordinal variables of the density of the collagen fibers (low, medium, high) according to standard guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontológica de la Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No